CLINICAL TRIAL: NCT01313234
Title: A Theory Based Educational Intervention Targeting Nurses Attitudes and Knowledge Concerning Cancer-related Pain Management: A Study Protocol of a Quasi-experimental Study Design
Brief Title: Educational Intervention Targeting Nurses Attitudes and Knowledge About Cancer-related Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BFR20100046019
Record Dates: First submitted 2011-03-05; First posted 2011-03-11 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Educational theory based intervention and systematic daily pain assessment
  Interventions: Behavioral: Education
- Control (No Intervention): Control group with care as usual

INTERVENTIONS:
Behavioral: Education — Theory based education and systematic daily assessment
  Arms: Education

SUMMARY:
The purpose of this study is to investigate whether an intervention consisting of the implementation of guidelines about daily systematic pain assessment following a theory based education, targeting cancer-related pain and pain treatment, lead to a significantly positive improvement in RNs knowledge of, and attitudes towards their pain management. Furthermore will the interventions targeting the RNs influence the admitted patient's perception of their cancer-related pain?

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Aged 18 years and above
* Cognitively intact and able to verbally communicate
* At admission pain intensity >1 on Visual Analogue Scale (VAS)

Exclusion Criteria:

* Trauma or planned and/or acute surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the total score of Knowledge and Attitudes Survey Regarding Pain | Measurement will occur at first session of the educational intervention and 2 and 6 weeks after
  Nurses attitude and knowledge as measured by a modified version of the instrument: Knowledge and Attitudes Survey Regarding Pain

SECONDARY OUTCOMES:
Change from Baseline - Brief Pain Inventory, Short Form (BPI-SF) | Measurement will occur at admission of the patient and at discharge from the hospital. Estimated average time period from admission to discharge is 2 weeks
  BPI-SF is a pain-assessment instrument developed for cancer patient. The instrument consists of nine items, and a figure depicting a human body where the patient marks position and type of pain. BPI-SF includes items concerning the degree of pain right now, pain during the last day and pain on average as well as items concerning effect of pain treatment, walking ability, mood, work, relationships and if sleep are affected by pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge Hospital, Karlskrona, Sweden

REFERENCES:
- [Derived] Gustafsson M, Borglin G. Can a theory-based educational intervention change nurses' knowledge and attitudes concerning cancer pain management? A quasi-experimental design. BMC Health Serv Res. 2013 Aug 19;13:328. doi: 10.1186/1472-6963-13-328. PMID 23958335
- [Derived] Borglin G, Gustafsson M, Krona H. A theory-based educational intervention targeting nurses' attitudes and knowledge concerning cancer-related pain management: a study protocol of a quasi-experimental design. BMC Health Serv Res. 2011 Sep 23;11:233. doi: 10.1186/1472-6963-11-233. PMID 21942991